CLINICAL TRIAL: NCT05895552
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of RTA 901 in Patients With Diabetic Peripheral Neuropathic Pain
Brief Title: A Study of RTA 901 (BIIB143) in Participants With Diabetic Peripheral Neuropathic Pain
Acronym: CYPRESS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to close study early; not due to safety concerns.
Sponsor: Reata, a wholly owned subsidiary of Biogen (Industry)
Responsible Party: Sponsor
Organization: Biogen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 297DP201; 901-C-2102 (Other: Reata, a wholly owned subsidiary of Biogen); NCT06893094 (obsolete NCT alias)
Record Dates: First submitted 2022-10-13; First posted 2023-06-08 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: RTA 901

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 RTA 901 Dose 1 (Experimental): Participants will receive study drug, once daily (QD), during the 2-week Run-in Period. Following randomization, the participants will receive a dose of RTA 901, QD, for a 12-week treatment duration.
  Interventions: Drug: RTA 901
- Part 1 RTA 901 Dose 2 (Experimental): Participants will receive study drug, QD, during the 2-week Run-in Period. Following randomization, the participants will receive a dose of RTA 901, QD, for a 12-week treatment duration.
  Interventions: Drug: RTA 901
- Part 1 RTA 901-Matching Placebo (Placebo Comparator): Participants will receive study drug, QD, during the 2-week Run-in Period. Following randomization, the participants will receive a dose of RTA 901-matching placebo, QD, for a 12-week treatment duration.
  Interventions: Drug: RTA 901-Matching Placebo
- Part 2 RTA 901 Dose 1 (Experimental): Participants will receive study drug, QD, during the 2-week Run-in Period. Following randomization, the participants will receive a dose of RTA 901, QD, for a 12-week treatment duration.
  Interventions: Drug: RTA 901
- Part 2 RTA 901 Dose 2 (Experimental): Participants will receive study drug, QD, during the 2-week Run-in Period. Following randomization, the participants will receive a dose of RTA 901, QD, for a 12-week treatment duration.
  Interventions: Drug: RTA 901
- Part 2 RTA 901-Matching Placebo (Placebo Comparator): Participants will receive study drug, QD, during the 2-week Run-in Period. Following randomization, the participants will receive a dose of RTA 901-matching placebo, QD, for a 12-week treatment duration.
  Interventions: Drug: RTA 901-Matching Placebo

INTERVENTIONS:
Drug: RTA 901 — Administered as specified in the treatment arm.
  Other Names: BIIB143; Cemdomespib
  Arms: Part 1 RTA 901 Dose 1; Part 1 RTA 901 Dose 2; Part 2 RTA 901 Dose 1; Part 2 RTA 901 Dose 2
Drug: RTA 901-Matching Placebo — Administered as specified in the treatment arm.
  Arms: Part 1 RTA 901-Matching Placebo; Part 2 RTA 901-Matching Placebo

SUMMARY:
This is a 2-part, randomized, placebo-controlled, double-blind, Phase 2 study to evaluate the safety, tolerability, efficacy, and pharmacokinetics (PK) of RTA 901 in qualified participants with Diabetic Peripheral Neuropathic Pain (DPNP). Each study part will be randomized into 3 treatment arms; 2 different doses of RTA 901 and RTA 901-maching placebo. The doses of RTA 901 in Part 2 will be selected based on the Exposure-Response (E-R) analyses of data from Part 1.

The duration of each part of the study will be approximately 20 weeks, including a Screening period of up to 2 weeks, a Run-in-period of 2 weeks, a Treatment period of 12 weeks, and a Follow-up period of 4 weeks. All participants in Part 1 and Part 2 of the study will follow the same visit and assessment schedule. Eligibility will be assessed during the Screening and Run-in-periods.

DETAILED DESCRIPTION:
Study Sponsor, originally Reata Pharmaceuticals, Inc., is now Reata Pharmaceuticals, Inc., a wholly owned subsidiary of Biogen.

ELIGIBILITY:
Run-in Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM) at least 1 year prior to Screening
* Clinical diagnosis of DPNP defined as symptomatic distal symmetric polyneuropathy (secondary to diabetes) in the lower extremities, which may include symptoms of pain that is burning, lancinating, tingling, or shooting (electric shock-like). Pain in the lower extremities may occur with paresthesia or dysesthesia (unpleasant sensations of burning). Neuropathic pain may be accompanied by an exaggerated response to painful stimuli (hyperalgesia) and pain evoked by light touch or contact, eg, with socks, shoes, and bedclothes (allodynia);
* NPRS pain intensity score ≥ 4 on an 11-point scale at Screening
* A score ≥ 2.5 on the Michigan Neuropathy Screening Instrument (MNSI) Part B

Run-in Exclusion Criteria:

* Has neuropathy from a cause other than T1DM or T2DM
* Has a condition other than DPNP that could confound the assessment of pain (eg, fibromyalgia or regional pain caused by lumbar or cervical compression);
* Diabetic foot ulceration or infection within 90 days prior to Screening
* Prior participation in a study with RTA 901;

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (75):
- United States (75):
  - Centricity Research Phoenix Multispecialty, Mesa, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Hope Clinical Research, Inc., Canoga Park, California
  - Valley Research - Trials, Fresno, California
  - Clinical Research Institute, Los Angeles, California
  - Acclaim Clinical Research, San Diego, California
  - Optimus Medical Group, San Francisco, California
  - PIH Health Whittier Hospital, Whittier, California
  - Denver Endocrinology Diabetes and Thyroid Center PC, Englewood, Colorado
  - Paradigm Clinical Research, Wheat Ridge, Colorado
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Clinical Research of West Florida Inc, Clearwater, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Multi Specialty Research Associates, LLC, Lake City, Florida
  - 3 Sync LLC, Lake Worth, Florida
  - Finlay Medical Research, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - IMA Clinical Research, PC, St. Petersburg, Florida
  - 3 Sync LLC, Sunrise, Florida
  - Genesis Clinical Research, Tampa, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Baycare Clinical Research, Tampa, Florida
  - VICIS Clinical Research, Tampa, Florida
  - Clinical Site Partners, Orlando, Winter Park, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - East Coast Institute for Research, LLC, Canton, Georgia
  - Centricity Research Columbus Endocrinology, Columbus, Georgia
  - East Coast Institute for Research, LLC, Macon, Georgia
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Tandem Clinical Research, Marrero, Louisiana
  - Tandem Clinical Research, Metairie, Louisiana
  - Boston Clinical Trials, LLC, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - ActivMed Practices & Research, LLC, Methuen, Massachusetts
  - Revival Research Institute, LLC., Sterling Heights, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Velocity Clinical Research, Inc., Lincoln, Nebraska
  - Velocity Clinical Research, Inc., Norfolk, Nebraska
  - Las Vegas Endocrinology, Henderson, Nevada
  - Jubilee Clinical Research Inc, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - ActivMed Practices & Research, LLC, Portsmouth, New Hampshire
  - Columbia University, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Carolina Institute for Clinical Research, LLC, Fayetteville, North Carolina
  - Diabetes & Endocrinology Associates of Stark County, Inc., Canton, Ohio
  - Velocity Clinical Research, Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Remington-Davis, Inc., Columbus, Ohio
  - Meta Medical Research Institute, Dayton, Ohio
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Notus Clinical Research, Charleston, South Carolina
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Trinity Clinical Research LLC, Tullahoma, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - REX Clinical Trials, LLC, Beaumont, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Care United Research, LLC, Forney, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Nerve and Muscle Center of Texas, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Endocrine IPS, PLLC, Houston, Texas
  - Amir A Hassan, MD, PA, Houston, Texas
  - 3 Sync LLC, Kingwood, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Shadow Creek Medical Clinic, Pearland, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at multiple investigative sites from 28 July 2023 to 15 November 2024.
Pre-assignment Details: This study was to be conducted in 2 parts: Part 1 to investigate the efficacy and safety of 10 milligrams (mg) and 80 mg doses of RTA 901 and Part 2 to investigate doses of RTA 901 between 1 mg and 80 mg once daily (QD) based on the exposure-response (E-R) analysis for efficacy in Part 1. The study was terminated after Part 1 was completed and did not proceed to Part 2. No participants were enrolled in Part 2.
Groups:
- Part 1: RTA 901 Matching Placebo + Standard-of-care (SOC): Participants received a single blind placebo, capsule, QD, orally, during the 2-week Run-in Period along with any one prescribed SOC pain medication (duloxetine, pregabalin, or gabapentin). Following randomization, the participants received a dose of RTA 901-matching placebo, QD, orally for 12-weeks during double blind treatment period.
- Part 1: RTA 901 10 mg + SOC: Participants received a single blind placebo, capsule, QD, orally, during the 2-week Run-in Period along with any one prescribed SOC pain medication (duloxetine, pregabalin, or gabapentin). Following randomization, the participants received RTA 901, 10 mg, QD, orally for 12-weeks during double blind treatment period.
- Part 1: RTA 901 80 mg + SOC: Participants received a single blind placebo, capsule, QD, orally, during the 2-week Run-in Period along with any one prescribed SOC pain medication (duloxetine, pregabalin, or gabapentin). Following randomization, the participants received RTA 901, 80 mg, QD, orally for 12-weeks during treatment period.
Period: Overall Study
Arm/Group | Part 1: RTA 901 Matching Placebo + Standard-of-care (SOC) | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Started | 69 | 70 | 70
Treated | 68 | 69 | 69
Completed | 65 | 63 | 62
Not Completed | 4 | 7 | 8
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Non-Compliance With Study Drug | 0 | 1 | 0
Not completed — Protocol Deviation | 0 | 0 | 2
Not completed — Failure to Meet Randomization Criteria | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) analysis set was defined as all randomized participants who received at least 1 dose of randomized study drug.
Groups:
- Part 1: RTA 901 Matching Placebo + SOC: Participants received a single blind placebo, capsule, QD, orally, during the 2-week Run-in Period along with any one prescribed SOC pain medication (duloxetine, pregabalin, or gabapentin). Following randomization, the participants received a dose of RTA 901-matching placebo, QD, orally for 12-weeks during double blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC | Total
Number analyzed (Participants) | 68 | 69 | 69 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (7.13) | 63.1 (9.97) | 64.6 (7.57) | 64.3 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 36 | 106
  Male | 31 | 36 | 33 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 31 | 34 | 33 | 98
  Ethnicity: Not Hispanic or Latino | 37 | 35 | 36 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 3 | 1 | 0 | 4
  Race: Black or African America | 14 | 16 | 15 | 45
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Race: White | 50 | 49 | 53 | 152
  Race: Multiple | 0 | 2 | 0 | 2
  Race: Other | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Average Pain Intensity Assessed by the Numeric Pain Rating Scale (NPRS) at Week 12
Description: The NPRS of pain intensity is an 11-point numeric scale, ranging from 0 (representing no pain at all) to 10 (representing the worst pain imaginable). The participants were asked to select a whole number (0 to 10) that best indicates the intensity of his/her neuropathic pain in the past 24 hours. The weekly average score of NPRS was defined as the sum of non-missing daily scores divided by the number of days with non-missing scores for that week. Negative change from baseline indicates decreased pain intensity.
Time Frame: Baseline, Week 12
Population: The ITT analysis set was defined as all randomized participants who received at least 1 dose of randomized study drug. Here, 'overall number of participants analyzed' signifies the number of participants evaluable for this outcome measure analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 65 | 63 | 63
score on a scale | -1.71 (0.249) | -1.49 (0.248) | -1.79 (0.248)
Statistical Analysis 1: Comparison: Part 1: RTA 901 Matching Placebo + SOC vs Part 1: RTA 901 10 mg + SOC; Test type: Superiority — The mixed model repeated measures (MMRM) model includes treatment group, baseline NPRS score, visit, interaction of visit and treatment group, and interaction of baseline NPRS score and visit; p < 0.5224, MMRM; Least square (LS) mean difference = 0.23, 95% CI 2-sided [-0.468 to 0.918], Standard Error of Mean 0.351
Statistical Analysis 2: Comparison: Part 1: RTA 901 Matching Placebo + SOC vs Part 1: RTA 901 80 mg + SOC; Test type: Superiority — The MMRM model includes treatment group, baseline NPRS score, visit, interaction of visit and treatment group, and interaction of baseline NPRS score and visit; p < 0.8223, MMRM; LS mean difference = -0.08, 95% CI 2-sided [-0.772 to 0.614], Standard Error of Mean 0.351

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) During and Following the Treatment Period
Description: An adverse event (AE) was any unfavorable and unintended sign (including any CS abnormal laboratory test result), symptom, or disease temporally associated with use of the study drug, whether or not it is considered to be study drug related. An SAE was any untoward medical occurrence that at any dose resulted in death, in the view of Investigator, placed participant at immediate risk of death, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in a birth defect. AEs that presented, or worsened in intensity or frequency, following the initiation of study treatment were categorized as TEAEs.
Time Frame: From the first dose of study drug up to end of follow-up period (up to 16 weeks)
Population: The safety analysis set includes all randomized participants who receive at least 1 dose of randomized study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 68 | 69 | 69
Participants
  TEAEs | 39 | 43 | 35
  SAEs | 4 | 5 | 1

3. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examinations
Description: Clinically significant abnormalities in physical examinations were based on investigator discretion.
Time Frame: From the first dose of study drug up to end of follow-up period (up to 16 weeks)
Population: The safety analysis set includes all randomized participants who received at least 1 dose of randomized study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 68 | 69 | 69
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Potential Clinically Significant Abnormalities in Vital Sign Parameters
Description: Vital sign parameters included temperature, pulse rate systolic blood pressure, diastolic blood pressure, and respiratory rate. As pre-specified in protocol, the criteria for determining potentially clinically relevant abnormalities in vital signs included: temperature < 36.0 and > 38.0 degrees Celsius (c), pulse rate < 60 and > 100 beats per minute (bpm), systolic blood pressure < 90, > 140 and > 160 millimeters of mercury (mmHg), diastolic blood pressure < 50, > 90 and > 100 mmHg, weight (7% or more increase from baseline, 7% or more decrease from baseline) and respiratory rate < 12 and > 20 breaths per minute. The categories with at least one participant with clinically significant vital sign abnormalities are reported.
Time Frame: From the first dose of study drug up to end of follow-up period (up to 16 weeks)
Population: The safety analysis set includes all randomized participants who received at least 1 dose of randomized study drug. Here, 'overall number of participants analyzed' signifies the number of participants evaluable for this outcome measure analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 67 | 69 | 68
Participants
  Temperature <36 degrees C | 15 | 17 | 16
  Temperature >38 degrees C | 0 | 1 | 0
  Pulse Rate <60 bpm | 18 | 6 | 11
  Pulse Rate >100 bpm | 3 | 1 | 1
  Systolic Blood Pressure <90 mmHg | 0 | 0 | 3
  Systolic Blood Pressure >140 mmHg | 24 | 28 | 22
  Systolic Blood Pressure >160 mmHg | 7 | 7 | 3
  Diastolic Blood Pressure <50 mmHg | 0 | 0 | 1
  Diastolic Blood Pressure >90 mmHg | 6 | 9 | 6
  Diastolic Blood Pressure >100 mmHg | 1 | 2 | 0
  Weight 7% or more increase from baseline | 1 | 1 | 2
  Weight 7% or more decrease from baseline | 1 | 1 | 1
  Respiratory Rate <12 breaths/min | 1 | 0 | 0
  Respiratory Rate >20 breaths/min | 1 | 1 | 1

5. Primary Outcome: Number of Participants With Shift From Baseline in Clinically Significant Abnormalities in Electrocardiogram (ECG)
Description: Clinical significance of abnormalities in ECG was determined based on the investigator's discretion.
Time Frame: From the first dose of study drug up to end of follow-up period (up to 16 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 27 | 34 | 30
Participants | 2 | 0 | 0

6. Primary Outcome: Number of Participants With Shift From Baseline in Clinical Laboratory Measurement (Hematology Parameters)
Description: Hematology parameters included hematocrit, hemoglobin, erythrocytes, leukocytes, neutrophils, lymphocytes, monocytes, basophils, eosinophils, platelets, mean corpuscular hemoglobin, mean corpuscular volume, and mean corpuscular hemoglobin concentration. These parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available. Here, shift to low indicated values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high postbaseline values. The categories with at least one participant with shift from baseline in these parameters are reported.
Time Frame: From the first dose of study drug up to end of follow-up period (up to 16 weeks)
Population: The safety analysis set includes all randomized participants who received at least 1 dose of randomized study drug. Here, 'overall number of participants analyzed' signifies the number of participants available for this outcome measure analysis. 'Number analyzed' signifies the number of participants with data available for analysis at specified time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 67 | 69 | 69
Participants
  Basophils/Leukocytes Shift to Low: number analyzed (Participants) | 67 | 69 | 68
  Basophils/Leukocytes Shift to Low | 0 | 0 | 0
  Basophils/Leukocytes Shift to High: number analyzed (Participants) | 67 | 69 | 68
  Basophils/Leukocytes Shift to High | 0 | 2 | 3
  Eosinophils Shift to Low: number analyzed (Participants) | 67 | 69 | 68
  Eosinophils Shift to Low | 0 | 0 | 0
  Eosinophils Shift to High: number analyzed (Participants) | 66 | 68 | 67
  Eosinophils Shift to High | 6 | 5 | 2
  Eosinophils/Leukocytes Shift to Low: number analyzed (Participants) | 67 | 69 | 68
  Eosinophils/Leukocytes Shift to Low | 0 | 0 | 0
  Eosinophils/Leukocytes Shift to High: number analyzed (Participants) | 58 | 63 | 66
  Eosinophils/Leukocytes Shift to High | 9 | 11 | 13
  Erythrocytes Mean Corpuscular Hemoglobin Concentration Shift to Low: number analyzed (Participants) | 58 | 61 | 62
  Erythrocytes Mean Corpuscular Hemoglobin Concentration Shift to Low | 19 | 19 | 23
  Erythrocytes Mean Corpuscular Hemoglobin Concentration Shift to High: number analyzed (Participants) | 67 | 69 | 68
  Erythrocytes Mean Corpuscular Hemoglobin Concentration Shift to High | 0 | 1 | 0
  Erythrocytes Mean Corpuscular Hemoglobin Shift to Low: number analyzed (Participants) | 62 | 63 | 63
  Erythrocytes Mean Corpuscular Hemoglobin Shift to Low | 3 | 0 | 4
  Erythrocytes Mean Corpuscular Hemoglobin Shift to High: number analyzed (Participants) | 66 | 68 | 68
  Erythrocytes Mean Corpuscular Hemoglobin Shift to High | 0 | 0 | 0
  Erythrocytes Mean Corpuscular Volume Shift to Low: number analyzed (Participants) | 62 | 65 | 61
  Erythrocytes Mean Corpuscular Volume Shift to Low | 2 | 2 | 1
  Erythrocytes Mean Corpuscular Volume Shift to High: number analyzed (Participants) | 67 | 69 | 67
  Erythrocytes Mean Corpuscular Volume Shift to High | 1 | 3 | 0
  Erythrocytes Shift to Low: number analyzed (Participants) | 63 | 58 | 60
  Erythrocytes Shift to Low | 7 | 6 | 10
  Erythrocytes Shift to High: number analyzed (Participants) | 64 | 64 | 67
  Erythrocytes Shift to High | 7 | 8 | 5
  Hematocrit Shift to Low: number analyzed (Participants) | 60 | 55 | 57
  Hematocrit Shift to Low | 14 | 7 | 12
  Hematocrit Shift to High: number analyzed (Participants) | 67 | 69 | 68
  Hematocrit Shift to High | 6 | 6 | 5
  Hemoglobin Shift to Low: number analyzed (Participants) | 62 | 57 | 58
  Hemoglobin Shift to Low | 11 | 8 | 13
  Hemoglobin Shift to High: number analyzed (Participants) | 66 | 67 | 67
  Hemoglobin Shift to High | 5 | 3 | 2
  Hemoglobin A1C/Hemoglobin Shift to Low: number analyzed (Participants) | 67 | 68 | 68
  Hemoglobin A1C/Hemoglobin Shift to Low | 0 | 0 | 0
  Hemoglobin A1C/Hemoglobin Shift to High: number analyzed (Participants) | 2 | 6 | 6
  Hemoglobin A1C/Hemoglobin Shift to High | 1 | 3 | 1
  Leukocytes Shift to Low: number analyzed (Participants) | 63 | 67 | 65
  Leukocytes Shift to Low | 4 | 7 | 11
  Leukocytes Shift to High: number analyzed (Participants) | 63 | 65 | 64
  Leukocytes Shift to High | 7 | 7 | 7
  Lymphocytes Shift to Low: number analyzed (Participants) | 62 | 69 | 67
  Lymphocytes Shift to Low | 3 | 2 | 4
  Lymphocytes Shift to High: number analyzed (Participants) | 66 | 69 | 68
  Lymphocytes Shift to High | 1 | 2 | 0
  Lymphocytes/Leukocytes Shift to Low: number analyzed (Participants) | 54 | 60 | 59
  Lymphocytes/Leukocytes Shift to Low | 15 | 23 | 17
  Lymphocytes/Leukocytes Shift to High: number analyzed (Participants) | 66 | 64 | 65
  Lymphocytes/Leukocytes Shift to High | 7 | 5 | 4
  Monocytes Shift to Low: number analyzed (Participants) | 67 | 69 | 68
  Monocytes Shift to Low | 0 | 0 | 0
  Monocytes Shift to High: number analyzed (Participants) | 65 | 66 | 66
  Monocytes Shift to High | 7 | 8 | 10
  Monocytes/Leukocytes Shift to Low: number analyzed (Participants) | 67 | 69 | 68
  Monocytes/Leukocytes Shift to Low | 0 | 2 | 0
  Monocytes/Leukocytes Shift to High: number analyzed (Participants) | 66 | 65 | 67
  Monocytes/Leukocytes Shift to High | 3 | 5 | 9
  Neutrophils Shift to Low: number analyzed (Participants) | 65 | 67 | 66
  Neutrophils Shift to Low | 1 | 1 | 3
  Neutrophils Shift to High: number analyzed (Participants) | 65 | 67 | 67
  Neutrophils Shift to High | 10 | 9 | 7
  Neutrophils/Leukocytes Shift to Low: number analyzed (Participants) | 67 | 65 | 68
  Neutrophils/Leukocytes Shift to Low | 2 | 4 | 3
  Neutrophils/Leukocytes Shift to High: number analyzed (Participants) | 56 | 65 | 61
  Neutrophils/Leukocytes Shift to High | 15 | 21 | 15
  Platelets Shift to Low: number analyzed (Participants) | 66 | 69 | 67
  Platelets Shift to Low | 2 | 0 | 1
  Platelets Shift to High: number analyzed (Participants) | 62 | 67 | 66
  Platelets Shift to High | 2 | 1 | 7

7. Primary Outcome: Number of Participants With Shift From Baseline in Clinical Laboratory Measurement (Blood Chemistry Parameters)
Description: Parameters included alanine aminotransferase (ALT), aspartate aminotransferase (AST), cholesterol, choriogonadotropin beta, follicle stimulating hormone (FSH), estimated glomerular filtration rate (eGFR), ferritin, creatine kinase, blood urea nitrogen, creatinine, bilirubin(total and direct), alkaline phosphatase, amylase, lipase, sodium, potassium, calcium, phosphorus, uric acid, total protein, glucose, albumin, lactate dehydrogenase, magnesium, chloride, bicarbonate, and gamma-glutamyl transferase. These parameters were flagged as low, normal or high relative to parameter's normal range or as unknown if no result was available, by Investigator. Here, shift to low indicates values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high values postbaseline. Categories with at least one participant with shift from baseline in these parameters are reported.
Time Frame: From the first dose of study drug up to end of follow-up period (up to 16 weeks)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 67 | 69 | 68
Participants
  ALT Shift to Low | 0 | 0 | 0
  ALT Shift to High: number analyzed (Participants) | 56 | 61 | 57
  ALT Shift to High | 13 | 17 | 13
  Albumin Shift to Low | 1 | 0 | 0
  Albumin Shift to High | 0 | 1 | 1
  Alkaline Phosphatase Shift to Low: number analyzed (Participants) | 62 | 66 | 68
  Alkaline Phosphatase Shift to Low | 2 | 3 | 1
  Alkaline Phosphatase Shift to High: number analyzed (Participants) | 54 | 56 | 51
  Alkaline Phosphatase Shift to High | 12 | 6 | 4
  Amylase Shift to Low: number analyzed (Participants) | 66 | 67 | 65
  Amylase Shift to Low | 1 | 2 | 2
  Amylase Shift to High: number analyzed (Participants) | 62 | 52 | 55
  Amylase Shift to High | 12 | 11 | 9
  AST Shift to Low: number analyzed (Participants) | 66 | 68 | 66
  AST Shift to Low | 9 | 7 | 5
  AST Shift to High: number analyzed (Participants) | 61 | 65 | 67
  AST Shift to High | 3 | 14 | 6
  Bicarbonate Shift to Low | 2 | 1 | 1
  Bicarbonate Shift to High: number analyzed (Participants) | 61 | 66 | 60
  Bicarbonate Shift to High | 5 | 9 | 5
  Bilirubin Shift to Low: number analyzed (Participants) | 65 | 67 | 67
  Bilirubin Shift to Low | 9 | 5 | 10
  Bilirubin Shift to High: number analyzed (Participants) | 66 | 68 | 64
  Bilirubin Shift to High | 1 | 3 | 2
  Calcium Shift to Low: number analyzed (Participants) | 66 | 68 | 65
  Calcium Shift to Low | 5 | 0 | 2
  Calcium Shift to High: number analyzed (Participants) | 67 | 66 | 64
  Calcium Shift to High | 6 | 2 | 8
  Chloride Shift to Low: number analyzed (Participants) | 62 | 69 | 66
  Chloride Shift to Low | 4 | 8 | 6
  Chloride Shift to High: number analyzed (Participants) | 66 | 68 | 65
  Chloride Shift to High | 6 | 7 | 5
  Cholesterol Shift to Low: number analyzed (Participants) | 67 | 68 | 68
  Cholesterol Shift to Low | 0 | 0 | 0
  Cholesterol Shift to High: number analyzed (Participants) | 57 | 57 | 60
  Cholesterol Shift to High | 9 | 6 | 11
  Creatine Kinase Shift to Low: number analyzed (Participants) | 63 | 67 | 65
  Creatine Kinase Shift to Low | 6 | 6 | 8
  Creatine Kinase Shift to High: number analyzed (Participants) | 60 | 52 | 55
  Creatine Kinase Shift to High | 17 | 23 | 18
  Creatinine Shift to Low: number analyzed (Participants) | 64 | 69 | 66
  Creatinine Shift to Low | 3 | 0 | 2
  Creatinine Shift to High: number analyzed (Participants) | 56 | 54 | 57
  Creatinine Shift to High | 16 | 11 | 15
  Direct Bilirubin Shift to Low | 0 | 0 | 0
  Direct Bilirubin Shift to High: number analyzed (Participants) | 65 | 64 | 62
  Direct Bilirubin Shift to High | 7 | 6 | 6
  Ferritin Shift to Low: number analyzed (Participants) | 57 | 60 | 58
  Ferritin Shift to Low | 9 | 6 | 10
  Ferritin Shift to High | 2 | 2 | 0
  Gamma Glutamyl Transferase Shift to Low | 0 | 0 | 0
  Gamma Glutamyl Transferase Shift to High: number analyzed (Participants) | 57 | 60 | 55
  Gamma Glutamyl Transferase Shift to High | 8 | 8 | 7
  eGFR Shift to Low: number analyzed (Participants) | 66 | 64 | 67
  eGFR Shift to Low | 14 | 10 | 12
  eGFR Shift to High | 0 | 0 | 0
  Glucose Shift to Low: number analyzed (Participants) | 66 | 69 | 67
  Glucose Shift to Low | 1 | 2 | 5
  Glucose Shift to High: number analyzed (Participants) | 14 | 17 | 19
  Glucose Shift to High | 14 | 14 | 16
  HDL Cholesterol Shift to Low: number analyzed (Participants) | 46 | 56 | 51
  HDL Cholesterol Shift to Low | 8 | 11 | 12
  HDL Cholesterol Shift to High: number analyzed (Participants) | 55 | 50 | 52
  HDL Cholesterol Shift to High | 3 | 6 | 3
  LDL Cholesterol Shift to Low: number analyzed (Participants) | 67 | 68 | 68
  LDL Cholesterol Shift to Low | 0 | 0 | 0
  LDL Cholesterol Shift to High: number analyzed (Participants) | 42 | 39 | 42
  LDL Cholesterol Shift to High | 11 | 10 | 11
  Lactate Dehydrogenase Shift to Low: number analyzed (Participants) | 64 | 69 | 67
  Lactate Dehydrogenase Shift to Low | 2 | 2 | 0
  Lactate Dehydrogenase Shift to High: number analyzed (Participants) | 66 | 64 | 67
  Lactate Dehydrogenase Shift to High | 5 | 10 | 11
  Lipase Shift to Low | 0 | 0 | 0
  Lipase Shift to High: number analyzed (Participants) | 42 | 46 | 51
  Lipase Shift to High | 17 | 22 | 23
  Magnesium Shift to Low: number analyzed (Participants) | 66 | 68 | 67
  Magnesium Shift to Low | 4 | 5 | 2
  Magnesium Shift to High: number analyzed (Participants) | 66 | 69 | 68
  Magnesium Shift to High | 1 | 1 | 2
  Phosphate Shift to Low: number analyzed (Participants) | 66 | 68 | 67
  Phosphate Shift to Low | 5 | 2 | 4
  Phosphate Shift to High: number analyzed (Participants) | 58 | 64 | 64
  Phosphate Shift to High | 14 | 21 | 16
  Potassium Shift to Low: number analyzed (Participants) | 66 | 69 | 67
  Potassium Shift to Low | 0 | 2 | 2
  Potassium Shift to High: number analyzed (Participants) | 60 | 59 | 62
  Potassium Shift to High | 19 | 22 | 20
  Protein Shift to Low: number analyzed (Participants) | 64 | 66 | 64
  Protein Shift to Low | 9 | 7 | 7
  Protein Shift to High: number analyzed (Participants) | 67 | 68 | 68
  Protein Shift to High | 1 | 0 | 0
  Sodium Shift to Low: number analyzed (Participants) | 65 | 69 | 68
  Sodium Shift to Low | 3 | 8 | 3
  Sodium Shift to High: number analyzed (Participants) | 63 | 64 | 66
  Sodium Shift to High | 8 | 8 | 7
  Triglycerides Shift to Low: number analyzed (Participants) | 67 | 68 | 68
  Triglycerides Shift to Low | 0 | 0 | 0
  Triglycerides Shift to High: number analyzed (Participants) | 41 | 48 | 45
  Triglycerides Shift to High | 17 | 16 | 21
  Urate Shift to Low: number analyzed (Participants) | 62 | 64 | 65
  Urate Shift to Low | 7 | 7 | 7
  Urate Shift to High: number analyzed (Participants) | 59 | 59 | 57
  Urate Shift to High | 11 | 9 | 11
  Urea Nitrogen Shift to Low: number analyzed (Participants) | 65 | 68 | 68
  Urea Nitrogen Shift to Low | 3 | 2 | 4
  Urea Nitrogen Shift to High: number analyzed (Participants) | 58 | 59 | 55
  Urea Nitrogen Shift to High | 14 | 23 | 15

8. Primary Outcome: Number of Participants With Shift From Baseline in Clinical Laboratory Measurement (Urinalysis)
Description: Urinalysis included assessments of bacteria, Bilirubin, Calcium Oxalate Crystals, Choriogonadotropin Beta, Color, Erythrocytes, Glucose, Granular Casts, Hyaline Casts, Ketones, Leukocyte Esterase, Leukocytes, Nitrite, Occult Blood, Protein, red blood cells (RBC) Casts, Renal Epithelial Cells, Specific Gravity, Specimen Appearance, Squamous Epithelial Cells, Transitional Epithelial Cells, Triple Phosphate Crystals, Uric Acid Crystals, white blood cells (WBC) Casts and pH. These parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available, by the Investigator. Here, shift to low indicates values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high postbaseline. The categories with at least one participant with shift from baseline in these parameters are reported.
Time Frame: From the first dose of study drug up to end of follow-up period (up to 16 weeks)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 67 | 69 | 68
Participants
  Bilirubin Shift to Low | 0 | 0 | 0
  Bilirubin Shift to High | 0 | 0 | 1
  Calcium Oxalate Crystals Shift to Low: number analyzed (Participants) | 52 | 49 | 50
  Calcium Oxalate Crystals Shift to Low | 0 | 0 | 0
  Calcium Oxalate Crystals Shift to High: number analyzed (Participants) | 50 | 43 | 46
  Calcium Oxalate Crystals Shift to High | 12 | 12 | 11
  Erythrocytes Shift to Low: number analyzed (Participants) | 52 | 49 | 50
  Erythrocytes Shift to Low | 0 | 0 | 0
  Erythrocytes Shift to High: number analyzed (Participants) | 51 | 46 | 47
  Erythrocytes Shift to High | 8 | 7 | 5
  Glucose Shift to Low | 0 | 0 | 0
  Glucose Shift to High: number analyzed (Participants) | 41 | 40 | 44
  Glucose Shift to High | 19 | 15 | 18
  Granular Casts Shift to Low: number analyzed (Participants) | 52 | 49 | 50
  Granular Casts Shift to Low | 0 | 0 | 0
  Granular Casts Shift to High: number analyzed (Participants) | 52 | 47 | 50
  Granular Casts Shift to High | 8 | 7 | 9
  Hyaline Casts Shift to Low: number analyzed (Participants) | 52 | 49 | 50
  Hyaline Casts Shift to Low | 0 | 0 | 0
  Hyaline Casts Shift to High: number analyzed (Participants) | 50 | 48 | 50
  Hyaline Casts Shift to High | 6 | 10 | 9
  Ketones Shift to Low | 0 | 0 | 0
  Ketones Shift to High: number analyzed (Participants) | 65 | 68 | 67
  Ketones Shift to High | 11 | 9 | 7
  Leukocyte Esterase Shift to Low | 0 | 0 | 0
  Leukocyte Esterase Shift to High: number analyzed (Participants) | 49 | 54 | 55
  Leukocyte Esterase Shift to High | 18 | 19 | 23
  Leukocytes Shift to Low: number analyzed (Participants) | 52 | 49 | 50
  Leukocytes Shift to Low | 0 | 0 | 0
  Leukocytes Shift to High: number analyzed (Participants) | 38 | 37 | 38
  Leukocytes Shift to High | 18 | 14 | 13
  Nitrite Shift to Low | 0 | 0 | 0
  Nitrite Shift to High: number analyzed (Participants) | 62 | 67 | 65
  Nitrite Shift to High | 5 | 7 | 7
  Occult Blood Shift to Low | 0 | 0 | 0
  Occult Blood Shift to High: number analyzed (Participants) | 65 | 66 | 65
  Occult Blood Shift to High | 15 | 10 | 5
  Protein Shift to Low | 0 | 0 | 0
  Protein Shift to High: number analyzed (Participants) | 57 | 53 | 53
  Protein Shift to High | 23 | 20 | 18
  RBC Casts Shift to Low: number analyzed (Participants) | 52 | 49 | 50
  RBC Casts Shift to Low | 0 | 0 | 0
  RBC Casts Shift to High: number analyzed (Participants) | 52 | 49 | 50
  RBC Casts Shift to High | 0 | 0 | 1
  Specific Gravity Shift to Low: number analyzed (Participants) | 64 | 68 | 66
  Specific Gravity Shift to Low | 8 | 11 | 12
  Specific Gravity Shift to High: number analyzed (Participants) | 55 | 58 | 55
  Specific Gravity Shift to High | 24 | 24 | 20
  Transitional Epithelial Cells Shift to Low: number analyzed (Participants) | 52 | 49 | 50
  Transitional Epithelial Cells Shift to Low | 3 | 0 | 0
  Transitional Epithelial Cells Shift to High: number analyzed (Participants) | 51 | 49 | 50
  Transitional Epithelial Cells Shift to High | 3 | 0 | 0
  Uric Acid Crystals Shift to Low: number analyzed (Participants) | 52 | 49 | 50
  Uric Acid Crystals Shift to Low | 0 | 0 | 0
  Uric Acid Crystals Shift to High: number analyzed (Participants) | 51 | 49 | 50
  Uric Acid Crystals Shift to High | 5 | 3 | 4
  WBC Casts Shift to Low: number analyzed (Participants) | 52 | 49 | 50
  WBC Casts Shift to Low | 0 | 0 | 0
  WBC Casts Shift to High: number analyzed (Participants) | 52 | 49 | 50
  WBC Casts Shift to High | 2 | 0 | 1
  Waxy Casts Shift to Low: number analyzed (Participants) | 52 | 49 | 50
  Waxy Casts Shift to Low | 0 | 0 | 0
  Waxy Casts Shift to High: number analyzed (Participants) | 52 | 49 | 50
  Waxy Casts Shift to High | 0 | 1 | 0
  Yeast Cells Shift to Low: number analyzed (Participants) | 52 | 49 | 50
  Yeast Cells Shift to Low | 0 | 0 | 0
  Yeast Cells Shift to High: number analyzed (Participants) | 52 | 48 | 48
  Yeast Cells Shift to High | 4 | 1 | 5
  pH Shift to Low | 0 | 0 | 0
  pH Shift to High: number analyzed (Participants) | 65 | 63 | 66
  pH Shift to High | 5 | 7 | 4

9. Primary Outcome: Number of Participants With Shift From Baseline in Clinical Laboratory Measurement (Coagulation Parameters)
Description: Coagulation included assessments of prothrombin. The parameter was flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available, by the Investigator. Here, shift to low indicates values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high postbaseline.
Time Frame: From the first dose of study drug up to end of follow-up period (up to 16 weeks)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 67 | 69 | 68
Participants
  Prothrombin International Normalized Ratio Shift to Low | 0 | 0 | 0
  Prothrombin International Normalized Ratio Shift to High: number analyzed (Participants) | 61 | 64 | 63
  Prothrombin International Normalized Ratio Shift to High | 13 | 20 | 16
  Prothrombin Time Shift to Low | 0 | 0 | 0
  Prothrombin Time Shift to High: number analyzed (Participants) | 57 | 62 | 62
  Prothrombin Time Shift to High | 14 | 21 | 19

10. Primary Outcome: Number of Participants With Clinically Significant Abnormality in Body Weight
Description: Weight decrease was characterized by a decrease of ≥7% from baseline and weight increase was characterized by an increase of ≥7% from baseline.
Time Frame: From the first dose of study drug up to end of follow-up period (up to 16 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 67 | 69 | 68
Participants
  Weight 7% or more increase from baseline | 1 | 1 | 2
  Weight 7% or more decrease from baseline | 1 | 1 | 1

11. Secondary Outcome: Number of Participants Who Achieved at Least a >=30% Decrease From Baseline in the Average NPRS Score at Week 12
Description: Responders is defined as participants with at least >=30% reduction in neuropathic pain from baseline in the NPRS average neuropathic pain intensity at Week 12 and were analysed using a logistic regression. The NPRS of pain intensity is a numeric scale, ranging from 0 (representing no pain at all) to 10 (representing the worst pain imaginable). The participant was asked to select a whole number (0 to 10) that best indicates the intensity of his/her neuropathic pain in the past 24 hours. Lower scores indicate less pain.
Time Frame: Baseline, Week 12
Population: The ITT analysis set was defined as all randomized participants who received at least 1 dose of randomized study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 68 | 69 | 69
Participants | 26 | 22 | 28

12. Secondary Outcome: Number of Participants Who Achieved at Least a >=50% Decrease From Baseline in the Average NPRS Score at Week 12
Description: Responder is defined as participants with at least >=50% reduction in neuropathic pain from baseline in the NPRS average neuropathic pain intensity at Week 12. The NPRS of pain intensity is a numeric scale, ranging from 0 (representing no pain at all) to 10 (representing the worst pain imaginable). The participant was asked to select a whole number (0 to 10) that best indicates the intensity of his/her neuropathic pain in the past 24 hours.
Time Frame: Baseline, Week 12
Population: The ITT analysis set was defined as all randomized participants who received at least 1 dose of randomized study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 68 | 69 | 69
Participants | 17 | 12 | 18

13. Secondary Outcome: Number of Participants Using Rescue Medications During the Treatment Period
Description: Rescue medication for diabetic peripheral neuropathic pain (DPNP) is in addition to standard of care medication (gabapentin, pregabalin or duloxetine) for DPNP. Rescue medication is intended to treat temporary elevations in a participant's DPNP and is intended to be used occasionally and not meant to be used for prolonged periods of time.
Time Frame: Up to Week 12
Population: The ITT analysis set was defined as all randomized participants who received at least 1 dose of randomized study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 68 | 69 | 69
Participants
  Week 1 | 20 | 15 | 22
  Week 2 | 19 | 16 | 19
  Week 3 | 20 | 15 | 22
  Week 4 | 18 | 13 | 18
  Week 5 | 15 | 11 | 18
  Week 6 | 14 | 10 | 16
  Week 7 | 10 | 14 | 16
  Week 8 | 14 | 14 | 19
  Week 9 | 11 | 10 | 13
  Week 10 | 7 | 10 | 15
  Week 11 | 9 | 10 | 12
  Week 12 | 10 | 13 | 14

14. Secondary Outcome: Amount of Rescue Medications Used During the Treatment Period
Description: The amount of rescue medication used per day during the 12-week treatment period was calculated as the total dosage recorded divided by total days of study drug exposure during the treatment period.
Time Frame: Up to Week 12
Population: The ITT analysis set was defined as all randomized participants who received at least 1 dose of randomized study drug.
Measure: Mean (Standard Deviation); unit: milligrams (mg) per day
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 68 | 69 | 69
milligrams (mg) per day
  NSAIDs | 18.40 (64.400) | 14.72 (51.060) | 48.15 (166.396)
  Acetaminophen | 55.50 (146.374) | 91.31 (308.725) | 101.09 (268.488)

15. Secondary Outcome: Time to First Occurrence of Rescue Medication Use
Description: Time to first occurrence of rescue medication use was defined as the time from first randomized dose to the first date of rescue medication use recorded in e-diary during the 12-week treatment period. If a participant withdraws from the study prior to week 12 and the participant did not take any rescue medication, then the participant will be censored on the last day in the study.
Time Frame: Up to Week 12
Population: The ITT analysis set was defined as all randomized participants who received at least 1 dose of randomized study drug. Here, 'overall number of participants analyzed' signifies the number of participants with first occurrence of rescue medication use.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 28 | 28 | 34
days | NA [16.0 to NA] — Median and upper values of 95% confidence interval were not estimable due to an insufficient number of participants with events. | NA [52.0 to NA] — Median and upper values of 95% confidence interval were not estimable due to an insufficient number of participants with events. | NA [15.0 to NA] — Median and upper values of 95% confidence interval were not estimable due to an insufficient number of participants with events.

16. Secondary Outcome: Change From Baseline in the Weekly Average of Daily Sleep Interference Scale (DSIS) Score at Week 12
Description: DSIS is a participant reported outcome that was developed to quantify sleep interference due to pain. The DSIS was completed daily by participants upon waking, preferably in the morning, to accurately capture variability in sleep interference due to pain, thus minimizing recall bias. Using the e-diary, participants assessed how neuropathic pain has interfered with their sleep during the past 24 hours. This score ranges from 0 to 10; 0 representing no interference with sleep to 10 representing complete inability to sleep, lower score indicating less pain interference during sleep. The weekly average score of DSIS was defined as the sum of non-missing daily scores divided by the number of days with non-missing scores for that week. A negative change from baseline indicates decreased interference in sleep due to pain.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 1: RTA 901 Matching Placebo + SOC | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
Number analyzed (Participants) | 66 | 63 | 63
score on a scale | -1.52 (2.035) | -1.41 (1.749) | -2.00 (2.249)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to end of follow-up period (Week 16)
Description: Adverse Events: The safety analysis set includes all randomized participants who received at least 1 dose of randomized study drug.
  All Cause Mortality: All randomized participants were included.
Groups:
- Part 1: RTA 901 Matching Placebo: Participants received a single blind placebo, capsule, QD, orally, during the 2-week Run-in Period along with any one prescribed SOC pain medication (duloxetine, pregabalin, or gabapentin). Following randomization, the participants received a dose of RTA 901-matching placebo, QD, orally for 12-weeks during double blind treatment period.
Arm/Group | Part 1: RTA 901 Matching Placebo | Part 1: RTA 901 10 mg + SOC | Part 1: RTA 901 80 mg + SOC
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 4/68 | 5/69 | 1/69
Other Adverse Events (participants affected / at risk) | 14/68 | 13/69 | 12/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: RTA 901 Matching Placebo (N=68) | Part 1: RTA 901 10 mg + SOC (N=69) | Part 1: RTA 901 80 mg + SOC (N=69)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: RTA 901 Matching Placebo (N=68) | Part 1: RTA 901 10 mg + SOC (N=69) | Part 1: RTA 901 80 mg + SOC (N=69)
Upper respiratory tract infection (Infections and infestations) | 5 | 1 | 3
Urinary tract infection (Infections and infestations) | 5 | 8 | 4
Blood creatine phosphokinase increased (Investigations) | 2 | 2 | 4
Lipase increased (Investigations) | 4 | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 5 | 2

LIMITATIONS AND CAVEATS:
The study was terminated prematurely based on the sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2024-05-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT05895552/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT05895552/SAP_001.pdf